CLINICAL TRIAL: NCT01276483
Title: Treatment Response Evaluation in Patients With Gastrointestinal Stromal Tumor Using PET/CT and DW MRI
Brief Title: Treatment Response Evaluation in Gastrointestinal Stromal Tumor (GIST) Patients
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mona-Elisabeth Revheim, Nuclear Medicine Phycisian, Oslo University Hospital
Other Study IDs: REK-2010/2089
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Soft Tissue Neoplasms; Gastrointestinal Tract
Keywords: GIST; Response Monitoring; Functional Magnetic Imaging; Positron Emission Tomography; Computer Tomography
MeSH Terms: conditions — Soft Tissue Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to compare sensitivity, specificity and accuracy of PET, DW MRI and CT separately and combined for the evaluation of treatment response and progression-free survival in patients with GIST.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic GIST patients suitable for TKI treatment
* GIST patients pursuing preoperative neoadjuvant TKI treatment

Exclusion Criteria:

* Patients with contraindications to MRI and/or TKI treatment. For patients with renal failure, CT without intravenous contrast will be performed according to clinical practice.
* Patients who do not sign the consent paper for any reason or do not accept the study premises or patients who wish to withdraw for any reason during the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: GIST patients suitable for medical treatment with targeted therapies.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-02; Primary Completion 2017-06 (Actual); Study Completion 2017-06-21 (Actual)

PRIMARY OUTCOMES:
Radiologic-pathologic correlation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mona-Elisabeth Revheim, MD, Principal Investigator — Oslo University Hospital, Dept of Nuclear Medicine; Therese Seierstad, PhD, Study Chair — Oslo University Hospital, Institute for Cancer Research; Øyvind S Bruland, Prof., MD, Principal Investigator — Oslo University Hospital, Dept of Oncology, The Norwegian Radium Hospital; Knut Håkon Hole, MD, Principal Investigator — Oslo University Hospital, Department of Diagnostic Radiology; Lars Julsrud, MD, Principal Investigator — Oslo University Hospital, Department of Diagnostic Radiology
Locations (1):
- Oslo University Hosptal, Oslo, Norway

REFERENCES:
- [Derived] Revheim ME, Hole KH, Bruland OS, Reitan E, Bjerkehagen B, Julsrud L, Seierstad T. Multimodal functional imaging for early response assessment in GIST patients treated with imatinib. Acta Oncol. 2014 Jan;53(1):143-8. doi: 10.3109/0284186X.2013.798428. Epub 2013 May 28. No abstract available. PMID 23710697